CLINICAL TRIAL: NCT01156571
Title: A Clinical Trial Comparing Cangrelor to Clopidogrel Standard of Care Therapy in Subjects Who Require Percutaneous Coronary Intervention (CHAMPION PHOENIX)
Brief Title: A Clinical Trial Comparing Cangrelor to Clopidogrel Standard Therapy in Subjects Who Require Percutaneous Coronary Intervention (PCI) (CHAMPION PHOENIX)
Acronym: CHAMPION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMC-CAN-10-01
Record Dates: First submitted 2010-06-29; First posted 2010-07-05 (Estimated); Results first posted 2013-06-18 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Atherosclerosis; Percutaneous Coronary Intervention; Acute Coronary Syndrome
MeSH Terms: conditions — Atherosclerosis; Acute Coronary Syndrome | interventions — Platelet Count; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- cangrelor (Experimental): Cangrelor was administered as a 30 µg/kg bolus followed by a 4.0 µg/kg/min cangrelor IV infusion for a minimum of 2 hours or until conclusion of the index procedure, whichever is longer. At the discretion of the treating physician, the infusion could be continued for a total duration of 4 hours.
  Following the discontinuation of the cangrelor infusion, 600mg of clopidogrel was administered.
  Interventions: Drug: cangrelor P2Y12 (platelet) inhibitor; Drug: Clopidogrel 600 mg post cangrelor
- clopidogrel (Active Comparator): Clopidogrel 300 mg or 600 mg administered pre or post PCI. Selection of dose and timing of dose were per investigator discretion.
  During the PCI a placebo infusion was given to maintain the blinding of the trial. In addition, placebo capsules were administered at the end of the infusion mimic the 600mg post infusion dose provided in the cangrelor arm.
  Interventions: Drug: Clopidogrel - 300 or 600 mg (study arm)

INTERVENTIONS:
Drug: cangrelor P2Y12 (platelet) inhibitor
  Arms: cangrelor
Drug: Clopidogrel - 300 or 600 mg (study arm) — Over encapsulated tablets.
  Arms: clopidogrel
Drug: Clopidogrel 600 mg post cangrelor — over-encapsulated clopidogrel (600 mg)
  Arms: cangrelor

SUMMARY:
The study is designed to compare the efficacy and safety profile of cangrelor to standard of care in patients require percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study if they meet all of the following criteria:

* Male or non-pregnant female at least 18 years of age
* Patients undergoing percutaneous coronary intervention (PCI):

  1. Stable angina (SA) patients with diagnostic coronary angiography within 90 days prior to randomization demonstrating atherosclerosis
  2. Non-ST-Segment Elevation Acute Coronary Syndrome (NSTE-ACS) patients with diagnostic coronary angiography within 72 hours prior to randomization demonstrating atherosclerosis
  3. ST-segment elevation myocardial infarction (STEMI) patients (diagnostic angiography not required)
* Provide written informed consent

Exclusion Criteria:

Patients will be excluded from the study if any of the following exclusion criteria apply prior to randomization:

* Receipt of any P2Y12 inhibitor at any time in the 7 days preceding randomization
* Eptifibatide and tirofiban usage within 12 hours preceding randomization (most recent dose must have been administered ≥12 hours prior to randomization)
* Abciximab usage within 7 days preceding randomization
* Receipt of fibrinolytic therapy in the 12 hours preceding randomization
* Increased bleeding risk: ischemic stroke within the last year or any previous hemorrhagic stroke; tumor, cerebral arteriovenous malformation, or intracranial aneurysm; recent (<1 month) trauma or major surgery (including bypass surgery); currently receiving warfarin; active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11145 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Anderson Area Medical Center, Anderson, South Carolina, United States

REFERENCES:
- [Derived] Gutierrez JA, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL; CHAMPION Investigators. Efficacy and safety of cangrelor in patients with peripheral artery disease undergoing percutaneous coronary intervention - Insights from the CHAMPION program. Am Heart J Plus. 2021 Aug 25;9:100043. doi: 10.1016/j.ahjo.2021.100043. eCollection 2021 Sep. PMID 38551015
- [Derived] Peterson BE, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL. Effect of Platelet Inhibition by Cangrelor Among Obese Patients Undergoing Coronary Stenting: Insights From CHAMPION. Circ Cardiovasc Interv. 2022 Mar;15(3):e011069. doi: 10.1161/CIRCINTERVENTIONS.121.011069. Epub 2022 Feb 24. PMID 35196863
- [Derived] Cavender MA, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Deliargyris EN, Prats J, Mahaffey KW, White HD, Bhatt DL; CHAMPION PHOENIX Investigators*. Ischemic Events Occur Early in Patients Undergoing Percutaneous Coronary Intervention and Are Reduced With Cangrelor: Findings From CHAMPION PHOENIX. Circ Cardiovasc Interv. 2022 Jan;15(1):e010390. doi: 10.1161/CIRCINTERVENTIONS.120.010390. Epub 2021 Dec 17. PMID 34915723
- [Derived] Olivier CB, Bhatt DL, Leonardi S, Stone GW, Gibson CM, Steg PG, Hamm CW, Wilson MD, Mangum S, Price MJ, Prats J, White HD, Lopes RD, Harrington RA, Mahaffey KW; CHAMPION PHOENIX Investigators *. Central Adjudication Identified Additional and Prognostically Important Myocardial Infarctions in Patients Undergoing Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2019 Jul;12(7):e007342. doi: 10.1161/CIRCINTERVENTIONS.118.007342. Epub 2019 Jul 12. PMID 31296081
- [Derived] Abtan J, Ducrocq G, Steg PG, Stone GW, Mahaffey KW, Gibson CM, Hamm CW, Price MJ, Prats J, Deliargyris EN, White HD, Harrington RA, Bhatt DL. Periprocedural Outcomes According to Timing of Clopidogrel Loading Dose in Patients Who Did Not Receive P2Y12 Inhibitor Pretreatment. Circ Cardiovasc Interv. 2019 Mar;12(3):e007445. doi: 10.1161/CIRCINTERVENTIONS.118.007445. PMID 30871355
- [Derived] Abtan J, Ducrocq G, Steg PG, Stone GW, Mahaffey KW, Gibson CM, Hamm C, Price MJ, Prats J, Elkin S, Deliargyris EN, White HD, Menozzi A, Harrington RA, Bhatt DL; MPH on Behalf of the CHAMPION PHOENIX Investigators. Characteristics and outcomes of patients requiring bailout use of glycoprotein IIb/IIIa inhibitors for thrombotic complications of percutaneous coronary intervention: An analysis from the CHAMPION PHOENIX trial. Int J Cardiol. 2019 Mar 1;278:217-222. doi: 10.1016/j.ijcard.2018.11.114. Epub 2018 Nov 23. PMID 30563770
- [Derived] Stone GW, Genereux P, Harrington RA, White HD, Gibson CM, Steg PG, Hamm CW, Mahaffey KW, Price MJ, Prats J, Deliargyris EN, Bhatt DL. Impact of lesion complexity on peri-procedural adverse events and the benefit of potent intravenous platelet adenosine diphosphate receptor inhibition after percutaneous coronary intervention: core laboratory analysis from 10 854 patients from the CHAMPION PHOENIX trial. Eur Heart J. 2018 Dec 7;39(46):4112-4121. doi: 10.1093/eurheartj/ehy562. PMID 30203006
- [Derived] Groves EM, Bhatt DL, Steg PG, Deliargyris EN, Stone GW, Gibson CM, Hamm CW, Mahaffey KW, White HD, Angiolillo DJ, Prats J, Harrington RA, Price MJ. Incidence, Predictors, and Outcomes of Acquired Thrombocytopenia After Percutaneous Coronary Intervention: A Pooled, Patient-Level Analysis of the CHAMPION Trials (Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition). Circ Cardiovasc Interv. 2018 Apr;11(4):e005635. doi: 10.1161/CIRCINTERVENTIONS.117.005635. PMID 29632238
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Steg G, Gibson CM, Hamm CW, Price MJ, Lopes RD, Leonardi S, Deliargyris EN, Prats J, Mahaffey KW, White HD, Bhatt DL. Short- and long-term mortality following bleeding events in patients undergoing percutaneous coronary intervention: insights from four validated bleeding scales in the CHAMPION trials. EuroIntervention. 2018 Feb 2;13(15):e1841-e1849. doi: 10.4244/EIJ-D-17-00723. PMID 28988157
- [Derived] Cavender MA, Bhatt DL, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Prats J, Elkin S, Deliargyris EN, Mahaffey KW, White HD, Harrington RA; CHAMPION PHOENIX Investigators*. Cangrelor in Older Patients Undergoing Percutaneous Coronary Intervention: Findings From CHAMPION PHOENIX. Circ Cardiovasc Interv. 2017 Aug;10(8):e005257. doi: 10.1161/CIRCINTERVENTIONS.117.005257. PMID 28801539
- [Derived] Parker WA, Bhatt DL, Prats J, Day JRS, Steg PG, Stone GW, Hamm CW, Mahaffey KW, Price MJ, Gibson CM, White HD, Storey RF; CHAMPION PHOENIX Investigators. Characteristics of dyspnoea and associated clinical outcomes in the CHAMPION PHOENIX study. Thromb Haemost. 2017 Jun 2;117(6):1093-1100. doi: 10.1160/TH16-12-0958. Epub 2017 Apr 6. PMID 28382371
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Deliargyris EN, Steg PG, Gibson CM, Hamm CW, Price MJ, Menozzi A, Prats J, Elkin S, Mahaffey KW, White HD, Bhatt DL; CHAMPION Investigators. Cangrelor With and Without Glycoprotein IIb/IIIa Inhibitors in Patients Undergoing Percutaneous Coronary Intervention. J Am Coll Cardiol. 2017 Jan 17;69(2):176-185. doi: 10.1016/j.jacc.2016.10.055. PMID 28081827
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Deliargyris EN, Steg PG, Gibson CM, Hamm CW, Price MJ, Menozzi A, Prats J, Elkin S, Mahaffey KW, White HD, Bhatt DL. Evaluation of Ischemic and Bleeding Risks Associated With 2 Parenteral Antiplatelet Strategies Comparing Cangrelor With Glycoprotein IIb/IIIa Inhibitors: An Exploratory Analysis From the CHAMPION Trials. JAMA Cardiol. 2017 Feb 1;2(2):127-135. doi: 10.1001/jamacardio.2016.4556. PMID 27902833
- [Derived] Abtan J, Steg PG, Stone GW, Mahaffey KW, Gibson CM, Hamm CW, Price MJ, Abnousi F, Prats J, Deliargyris EN, White HD, Harrington RA, Bhatt DL; CHAMPION PHOENIX Investigators. Efficacy and Safety of Cangrelor in Preventing Periprocedural Complications in Patients With Stable Angina and Acute Coronary Syndromes Undergoing Percutaneous Coronary Intervention: The CHAMPION PHOENIX Trial. JACC Cardiovasc Interv. 2016 Sep 26;9(18):1905-13. doi: 10.1016/j.jcin.2016.06.046. PMID 27659566
- [Derived] Cavender MA, Bhatt DL, Stone GW, White HD, Steg PG, Gibson CM, Hamm CW, Price MJ, Leonardi S, Prats J, Deliargyris EN, Mahaffey KW, Harrington RA; CHAMPION PHOENIX Investigators*. Consistent Reduction in Periprocedural Myocardial Infarction With Cangrelor as Assessed by Multiple Definitions: Findings From CHAMPION PHOENIX (Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition). Circulation. 2016 Sep 6;134(10):723-33. doi: 10.1161/CIRCULATIONAHA.115.020829. Epub 2016 Aug 1. PMID 27482008
- [Derived] Vaduganathan M, Harrington RA, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL. Variation in Patient Profiles and Outcomes in US and Non-US Subgroups of the Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition (CHAMPION) PHOENIX Trial. Circ Cardiovasc Interv. 2016 Jun;9(6):e003612. doi: 10.1161/CIRCINTERVENTIONS.116.003612. PMID 27313282
- [Derived] O'Donoghue ML, Bhatt DL, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Prats J, Liu T, Deliargyris EN, Mahaffey KW, White HD, Harrington RA; CHAMPION PHOENIX Investigators. Efficacy and Safety of Cangrelor in Women Versus Men During Percutaneous Coronary Intervention: Insights From the Cangrelor versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition (CHAMPION PHOENIX) Trial. Circulation. 2016 Jan 19;133(3):248-55. doi: 10.1161/CIRCULATIONAHA.115.017300. PMID 26762525
- [Derived] Gutierrez JA, Harrington RA, Blankenship JC, Stone GW, Steg PG, Gibson CM, Hamm CW, Price MJ, Genereux P, Prats J, Deliargyris EN, Mahaffey KW, White HD, Bhatt DL; CHAMPION PHOENIX Investigators. The effect of cangrelor and access site on ischaemic and bleeding events: insights from CHAMPION PHOENIX. Eur Heart J. 2016 Apr 7;37(14):1122-30. doi: 10.1093/eurheartj/ehv498. Epub 2015 Sep 23. PMID 26400827
- [Derived] Genereux P, Stone GW, Harrington RA, Gibson CM, Steg PG, Brener SJ, Angiolillo DJ, Price MJ, Prats J, LaSalle L, Liu T, Todd M, Skerjanec S, Hamm CW, Mahaffey KW, White HD, Bhatt DL; CHAMPION PHOENIX Investigators. Impact of intraprocedural stent thrombosis during percutaneous coronary intervention: insights from the CHAMPION PHOENIX Trial (Clinical Trial Comparing Cangrelor to Clopidogrel Standard of Care Therapy in Subjects Who Require Percutaneous Coronary Intervention). J Am Coll Cardiol. 2014 Feb 25;63(7):619-629. doi: 10.1016/j.jacc.2013.10.022. Epub 2013 Oct 30. PMID 24184169
- [Derived] Bhatt DL, Stone GW, Mahaffey KW, Gibson CM, Steg PG, Hamm CW, Price MJ, Leonardi S, Gallup D, Bramucci E, Radke PW, Widimsky P, Tousek F, Tauth J, Spriggs D, McLaurin BT, Angiolillo DJ, Genereux P, Liu T, Prats J, Todd M, Skerjanec S, White HD, Harrington RA; CHAMPION PHOENIX Investigators. Effect of platelet inhibition with cangrelor during PCI on ischemic events. N Engl J Med. 2013 Apr 4;368(14):1303-13. doi: 10.1056/NEJMoa1300815. Epub 2013 Mar 10. PMID 23473369
- [Derived] Leonardi S, Mahaffey KW, White HD, Gibson CM, Stone GW, Steg GW, Hamm CW, Price MJ, Todd M, Dietrich M, Gallup D, Liu T, Skerjanec S, Harrington RA, Bhatt DL. Rationale and design of the Cangrelor versus standard therapy to acHieve optimal Management of Platelet InhibitiON PHOENIX trial. Am Heart J. 2012 May;163(5):768-776.e2. doi: 10.1016/j.ahj.2012.02.018. PMID 22607853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date first patient enrolled: 30 Sep 2010 Date last patient completed: 14 Nov 2012
  This trial enrolled the full spectrum of patients who required PCI (SA, NSTE-ACS, STEMI). Randomization occurred after confirmation of need for PCI (after diagnostic angiogram in all cases, except for STEMI patients). Patients were followed through 30-days.
Pre-assignment Details: Due to the nature of the disease, STEMI patients were permitted to be randomized upon ECG confirmation and prior to confirmation of need for PCI (prior to diagnostic angiography). Therefore in some cases, STEMI patients did not require PCI and therefore did not receive all study drug.
Groups:
- Cangrelor Treatment Arm: Cangrelor was administered as a 30 µg/kg bolus followed by a 4.0 µg/kg/min cangrelor IV infusion for a minimum of 2 hours or until conclusion of the index procedure, whichever is longer. At the discretion of the treating physician, the infusion could be continued for a total duration of 4 hours.
  Immediately after discontinuation of infusion, an oral transition dose of clopidogrel 600 mg was administered.
  Patients also received oral placebo capsules, administered as soon as possible following randomization at investigator discretion. These capsules were designed to match the clopidogrel 600 mg or 300 mg loading dose.
- Clopidogrel Treatment Arm: Oral clopidogrel was administered as soon as possible following randomization at investigator discretion at a loading dose of either 600 mg or 300 mg as specified by the investigator.
  Patients in the clopidogrel treatment arm received IV placebo for 2 hours or end of the PCI procedure, whichever was longer. At the discretion of the treating physician, the infusion could be continued for a total duration of 4 hours.
  At the end of IV placebo infusion, patients were given oral placebo capsules matching the oral clopidogrel transition dose.
Period: Overall Study
Arm/Group | Cangrelor Treatment Arm | Clopidogrel Treatment Arm
Started | 5581 (ITT: defined as all patients randomized.) | 5564 (ITT: defined as all patients randomized.)
Completed | 5564 (Completed = ITT patients who completed scheduled visits or developed a primary endpoint event) | 5545 (Completed = ITT patients who completed scheduled visits or developed a primary endpoint event)
Not Completed | 17 | 19

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cangrelor Treatment Arm | Clopidogrel Treatment Arm | Total
Number analyzed (Participants) | 5581 | 5564 | 11145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2892 | 2902 | 5794
  >=65 years | 2689 | 2662 | 5351
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (11.0) | 63.8 (11.0) | 63.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1599 | 1522 | 3121
  Male | 3982 | 4042 | 8024
Region of Enrollment [Number; unit: participants]
  United States | 2099 | 2089 | 4188
  Austria | 302 | 300 | 602
  Brazil | 78 | 80 | 158
  Bulgaria | 169 | 167 | 336
  Czech Republic | 814 | 816 | 1630
  Georgia | 744 | 741 | 1485
  Germany | 243 | 251 | 494
  Italy | 311 | 310 | 621
  New Zealand | 22 | 23 | 45
  Poland | 352 | 350 | 702
  Russian Federation | 296 | 286 | 582
  Thailand | 151 | 151 | 302

OUTCOME MEASURES:

1. Primary Outcome: The Composite Incidence of All-cause Mortality, Myocardial Infarction (MI), Ischemia-driven Revascularization (IDR) and Stent Thrombosis (ST)
Description: Clinical Events Committee (CEC)-adjudicated results (modified intent-to-treat [mITT] population)
Time Frame: 48 hours after randomization
Measure: Number; unit: participants
Arm/Group | Cangrelor Treatment Arm | Clopidogrel Treatment Arm
Number analyzed (Participants) | 5470 | 5469
participants | 257 | 322

2. Secondary Outcome: Individual Incidence of Stent Thrombosis (ST), Death, Myocardial Infarction (MI) and Ischemia-driven Revascularization (IDR)
Description: CEC-adjudicated results (mITT population)
Time Frame: 48 hours after randomization
Measure: Number; unit: participants
Arm/Group | Cangrelor Treatment Arm | Clopidogrel Treatment Arm
Number analyzed (Participants) | 5470 | 5469
participants
  Stent Thrombosis | 46 | 74
  Death | 18 | 18
  MI (myocardial infarction) | 207 | 255
  IDR (ischemia-driven revascularization) | 28 | 38

3. Secondary Outcome: Incidence of Major/Minor Non-coronary Artery Bypass Graft (CABG)-Related Hemorrhage by Clinical Relevant Criteria - GUSTO Severe/Life-threatening, Moderate and Mild
Description: GUSTO = Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries trial
Time Frame: 48 hours after randomization
Measure: Number; unit: participants
Arm/Group | Cangrelor Treatment Arm | Clopidogrel Treatment Arm
Number analyzed (Participants) | 5529 | 5527
participants
  GUSTO severe/life threatening | 9 | 6
  GUSTO moderate | 22 | 13
  GUSTO severe or moderate | 31 | 19
  TIMI major | 5 | 5
  TIMI minor | 9 | 3
  TIMI major or minor | 14 | 8
  Any blood transfusion | 25 | 16

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of randomization until 48 hours after randomization. If there was a delay between randomization and study drug initiation, AEs were collected from randomization through 48 hours after study drug initiation.
Arm/Group | Cangrelor Treatment Arm | Clopidogrel Treatment Arm
Serious Adverse Events (participants affected / at risk) | 122/5529 | 105/5527
Other Adverse Events (participants affected / at risk) | 0/5529 | 0/5527
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cangrelor Treatment Arm (N=5529) | Clopidogrel Treatment Arm (N=5527)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypersplenism (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
acute coronary syndrome (Cardiac disorders) | 1 | 0
acute myocardial infarction (Cardiac disorders) | 2 | 3
angina pectoris (Cardiac disorders) | 1 | 1
angina unstable (Cardiac disorders) | 2 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 0
atrial fibrillation (Cardiac disorders) | 2 | 2
atrioventricular block complete (Cardiac disorders) | 3 | 3
bradycardia (Cardiac disorders) | 1 | 1
cardiac arrest (Cardiac disorders) | 5 | 8
cardiac failure (Cardiac disorders) | 1 | 3
cardiac failure acute (Cardiac disorders) | 1 | 0
cardiac failure congestive (Cardiac disorders) | 3 | 3
cardiac tamponade (Cardiac disorders) | 1 | 0
cardio-respiratory arrest (Cardiac disorders) | 3 | 1
cardiogenic shock (Cardiac disorders) | 12 | 6
coronary artery disease (Cardiac disorders) | 0 | 1
coronary artery dissection (Cardiac disorders) | 9 | 6
coronary artery occlusion (Cardiac disorders) | 0 | 4
coronary artery performation (Cardiac disorders) | 3 | 3
Interventricluar septum rupture (Cardiac disorders) | 2 | 0
myocardial infarction (Cardiac disorders) | 2 | 1
mycardial rupture (Cardiac disorders) | 0 | 3
nodal arrhythmia (Cardiac disorders) | 1 | 1
percarditis (Cardiac disorders) | 0 | 1
sick sinus syndrome (Cardiac disorders) | 1 | 1
sinus arrest (Cardiac disorders) | 1 | 0
ventricular rupture (Cardiac disorders) | 1 | 0
ventricular asystole (Cardiac disorders) | 0 | 1
ventricular fibrillation (Cardiac disorders) | 6 | 7
ventricluar tachycardia (Cardiac disorders) | 5 | 3
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
chest discomfort (General disorders) | 1 | 0
chest pain (General disorders) | 5 | 2
non-cardiac chest pain (General disorders) | 2 | 0
pyrexia (General disorders) | 0 | 1
thrombosis in device (General disorders) | 3 | 3
hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
anaphylactic reaction (Immune system disorders) | 2 | 0
anaphylactic shock (Immune system disorders) | 1 | 0
hypersensitivity (Immune system disorders) | 0 | 2
bronchitis (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 1 | 1
septic shock (Infections and infestations) | 1 | 0
small intestine gangrene (Infections and infestations) | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 1
cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
fall (Injury, poisoning and procedural complications) | 0 | 1
head injury (Injury, poisoning and procedural complications) | 0 | 1
medication error (Injury, poisoning and procedural complications) | 1 | 0
postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
blood creatinine increased (Investigations) | 3 | 1
electrocardiogram ST segment elevation (Investigations) | 0 | 1
troponin increased (Investigations) | 1 | 2
diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
fluid overload (Metabolism and nutrition disorders) | 0 | 1
compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
cerebrovascular accident (Nervous system disorders) | 0 | 2
embolic cerebral infarction (Nervous system disorders) | 0 | 1
ischaemic stroke (Nervous system disorders) | 2 | 1
lethargy (Nervous system disorders) | 0 | 1
migraine (Nervous system disorders) | 1 | 0
presyncope (Nervous system disorders) | 1 | 3
transient ischaemic attack (Nervous system disorders) | 1 | 1
delirium (Psychiatric disorders) | 1 | 1
mental status changes (Psychiatric disorders) | 0 | 3
nephrolithiasis (Renal and urinary disorders) | 1 | 0
nephropathy toxic (Renal and urinary disorders) | 1 | 2
renal failure (Renal and urinary disorders) | 2 | 1
renal failure acute (Renal and urinary disorders) | 2 | 2
renal impairment (Renal and urinary disorders) | 1 | 0
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 3
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
aortic dissection (Vascular disorders) | 1 | 0
arterial rupture (Vascular disorders) | 2 | 2
circulatory collapse (Vascular disorders) | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 0
hypertension (Vascular disorders) | 0 | 1
hypotension (Vascular disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, PI communications regarding trial results are prohibited until after the communication and publication of the multi-center results by Sponsor, but no more than 12 months after conclusion of the trial at all sites.

PI must submit results communications to sponsor for review at least 45 days prior to submission for publication and Sponsor may embargo such communications for a period that is less than or equal to 135 days solely to seek appropriate patent protection.